CLINICAL TRIAL: NCT03882931
Title: Functional Roles of Dorsolateral Prefrontal Cortex in Visuomotor Adaptation and Response Selection
Brief Title: Functional Roles of Dorsolateral Prefrontal Cortex
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Virginia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 21068
Record Dates: First submitted 2019-03-19; First posted 2019-03-20 (Actual); Last update posted 2019-11-19 (Actual); Status verified 2019-11

CONDITIONS: Healthy Participants
Keywords: Dorsolateral Prefrontal Cortex; Neuromodulation; Transcranial Magnetic Stimulation; Transcranial Ultrasound Stimulation
MeSH Terms: interventions — salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants receiving ultrasound stimulation will be blinded to the type of ultrasound stimulation they are receiving.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- TMS to left DLPFC (Experimental): Theta Burst Transcranial Magnetic Stimulation will be delivered at 80% of the participants motor threshold to the left DLPFC and complete a visuomotor rotation task.
  Interventions: Other: Theta Burst Transcranial Magnetic Stimulation
- TMS to right DLPFC (Experimental): Theta Burst Transcranial Magnetic Stimulation will be delivered at 80% of the participants motor threshold to the right DLPFC and complete a visuomotor rotation task.
  Interventions: Other: Theta Burst Transcranial Magnetic Stimulation
- TMS Control (Sham Comparator): A Sham Theta Burst Transcranial Magnetic Stimulation will be delivered to the right/left DLPFC and complete a visuomotor rotation task.
  Interventions: Other: Sham
- FUS to right/left DLPFC (Experimental): Low intensity Focused Ultrasound stimulation will be delivered to either the left or right DLPFC depending on the subject's DLPFC response during their functional MRI flanker task.
  Interventions: Other: Focused Ultrasound

INTERVENTIONS:
Other: Theta Burst Transcranial Magnetic Stimulation — Theta Bursts are short bursts of stimulation at high frequencies, which are applied 5 times per second
  Arms: TMS to left DLPFC; TMS to right DLPFC
Other: Focused Ultrasound — Low intensity focused ultrasound is sound energy stimulation at a low intensity of 1-30 W/cm2
  Arms: FUS to right/left DLPFC
Other: Sham — The investigators will simulate theta bursts pulses similar to the Theta Burst Transcranial Magnetic Stimulation groups but without stimulation.
  Arms: TMS Control

SUMMARY:
Dorsolateral prefrontal cortex (DLPFC) has been found to be involved in cognitive functions such as executive function, response selection, and working memory. By applying transcranial magnetic stimulation (TMS) or transcranial focused ultrasound (FUS), which is a technology to temporally alter brain state in the stimulation site, the investigators aim to find supporting evidence for the causal relationship between the targeted stimulation site and motor learning improvement or response selection.

DETAILED DESCRIPTION:
The purpose of this study is to test the functions of dorsolateral prefrontal cortex in human motor learning. Dorsolateral prefrontal cortex (DLPFC) has been found to be involved in cognitive functions such as executive function, response selection, and working memory. Recent Findings hint potential involvement of dorsolateral prefrontal cortex in motor learning. Rare studies provided supporting evidence on its involvement and functions. This study aims to examine the functional roles of dorsolateral prefrontal cortex in human motor learning. By applying transcranial magnetic stimulation (TMS) or transcranial focused ultrasound (FUS), which is a technology to temporally alter brain state in the stimulation site, the investigators aim to find supporting evidence for the causal relationship between the targeted stimulation site and motor learning improvement or response selection.

Young healthy adults will be recruited and randomly assigned to one of four experimental groups. If randomized into one of the TMS groups, participants will learn to adapt to two visual rotations (20 and 60 degrees) when reaching for a virtual target, subjects will receive repetitive TMS (rTMS) stimulation over the targeted location, left DLPFC, or right DLPFC depending on the study group. How rTMS stimulation influencing the acquisition and retention of motor memory will be assessed based on group comparison of behavioral measures such as reaching accuracy. If randomized into the FUS group, participants will complete a flanker task to focuses on the assessment of response selection and inhibitory control.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, adult subjects
* 18 to 35 years of age
* Right-handed
* Have no any type of metal in the body
* Provide written informed consent

Exclusion Criteria:

* Presence of a significant medical, psychiatric, or neurologic illness
* History of loss of consciousness of more than ten minutes in the past year or loss of consciousness in a lifetime that required rehabilitation services
* Personal or family history of seizure
* Any history of stroke/transient ischemic attack (TIA) or severe traumatic brain injury
* Taking any medications that may decrease the threshold for seizure
* Pregnancy (self-reported)
* Affirmative answers to one or more questions of the provided attached safety questionnaires. These are not absolute contraindications to this study but the risk/benefit ratio will be carefully balanced by the PI
* Failure to follow laboratory or study procedures

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2019-01-28 (Actual); Primary Completion 2020-01-27 (Estimated); Study Completion 2020-01-27 (Estimated)

PRIMARY OUTCOMES:
Performance Error on Visuomotor Task | immediately following baseline assessment
  The visuomotor task has practice, baseline, and experimental trials. Performance on the task will be compared between groups.

CONTACTS AND LOCATIONS:
Overall Officials: Wynn Legon, PhD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: Undecided